# STATISTICAL ANALYSIS PLAN

Final Version 2.0 18/02/2019

OTIVACTO (1237.58)

Assessment of physical functioning and handling of Spiolto® Respimat® in patients with chronic obstructive pulmonary disease (COPD) requiring long-acting dual bronchodilation in routine clinical practice

**Sponsor** 



Document:

OTIVACTO - SAP\_v 2 0\_20190218

# **SIGNATURE SHEET**

| | Person responsible | Signature | Date<br>(dd/mm/yyyy) |
|--------------|---------------------|-----------|----------------------|
| Prepared by: | Statistician | | |
| Reviewed by: | Statistician 2 | | |
| neviewed by. | Project | | |
| Approved by: | Global Statistician | | |
| | Sponsor Project | | |

1. GENERAL INFORMATION ABOUT THE STUDY

1.1. Sponsor identification

Boehringer Ingelheim España, S.A.

C/ Prat de la Riba, 50

08174 Sant Cugat del Vallès (Barcelona)

1.2. STUDY TITLE

Assessment of physical functioning and handling of Spiolto® Respimat® in patients with chronic

obstructive pulmonary disease (COPD) requiring long-acting dual bronchodilation in routine

clinical practice

**1.3.** Protocol code

BI study number: 1237.58

1.4. COORDINATING INVESTIGATOR/S

1.5. Types of site where the study will be conducted

It is expected that data will be collected from approximately 200 sites (primary care centres)

in Spain. Sites will be selected in a way that reflects routine clinical practice for COPD in order

to ensure the representativeness of the population with COPD. The inclusion of 5 patients

per investigator has been planned.

1.6. IEC EVALUATING THE STUDY

Badajoz IEC, in Spain

1.7. PRIMARY OBJECTIVE

The primary objective of the study is to measure changes in physical functioning - serving as a

surrogate for physical activity and exercise capacity - in COPD patients being treated with


Spiolto® Respimat® after approximately 6 weeks.

1.8. STUDY DESIGN

This is an observational study, since the pharmaceutical product is prescribed in accordance

with routine clinical practice. The allocation of the patient to a particular therapeutic strategy

is not decided in advance in the study protocol, but it will be determined by routine clinical

practice and the decision to prescribe a specific medicinal product will be clearly disassociated

from the decision to include the patient in the study. No other clinical intervention (or

diagnosis, or clinical follow-up) which is different from routine clinical practice will be

applicable in the study.

This is a self-controlled study design which will include patients with COPD who have given

their consent and who will be treated with Spiolto® Respimat® in accordance with the

product's authorised summary of product characteristics.

Patients will be included consecutively and follow-up will be carried out over an observation

period of approximately 6 weeks.

The decision to treat with Spiolto® Respimat® will be taken independently of the participation

in this NIS and will be made before participation is considered.

1.9. DISEASE(S) OR DISORDER(S) UNDER STUDY

Chronic obstructive pulmonary disease (COPD)

1.10. Information on the study medicinal products

Spiolto® Respimat® 2.5 micrograms/2.5 micrograms solution for inhalation;

tiotropium/olodaterol

1.11. STUDY POPULATION AND TOTAL NUMBER OF SUBJECTS

COPD patients requiring a fixed combination therapy of two long-acting bronchodilators

(LAMA + LABA) according to approved SmPC and GOLD guidelines. Approximately 1000


patients will be included.

1.12.STUDY SCHEDULE

The planned schedule is as follows:

| Milestone | Planned date |
|---------------------------------|------------------------|
| Start of data collection (FPFV) | 24/04/2017 |
| End of data collection (LPLV) | 18/09/2018 (estimated) |
| Final report of study results | June 2019 (estimated) |

FPFV: First Patient First Visit; LPLV: Last Patient Last Visit

# 1.13. SOURCE OF FUNDING

Boehringer Ingelheim España, S.A. C/ Prat de la Riba, 50 08174 Sant Cugat del Vallès (Barcelona)

# 1.14. DETAILS OF THE COORDINATING SITE

Tel.: Fax:

OTIVACTO (1237.58) - SAP Date: 18/02/2019 (Final Version 2.0)

# **CONTENTS**

| 1. | GENE | RAL INFORMATION ABOUT THE STUDY | 3 |
|----|------|-----------------------------------------------------------|----|
| 2. | GLOS | SARY OF ABBREVIATIONS | 12 |
| 3. | STUD | Y OBJECTIVES | 13 |
| | 3.1. | PRIMARY OBJECTIVE | 13 |
| | 3.2. | SECONDARY OBJECTIVES | 13 |
| 4. | STUD | Y POPULATION | 14 |
| | 4.1. | Selection criteria | 14 |
| | | 4.1.1. Inclusion criteria | 14 |
| | | 4.1.2. Exclusion criteria | 14 |
| | 4.2. | RATIONALE FOR SAMPLE SIZE | 15 |
| 5. | METH | HODS | 16 |
| | 5.1. | Data processing | 16 |
| | 5.2. | DATA ANALYSIS AND STATISTICAL TESTS | 16 |
| | | 5.2.1. Important protocol violations | 16 |
| | | 5.2.2. Population for analysis | 17 |
| | | 5.2.3. Analysis of primary endpoint | 17 |
| | | 5.2.4. Analysis of secondary endpoints | 17 |
| | | 5.2.5. Analysis of other endpoints | 18 |
| | | 5.2.7. Statistical methodology | 21 |
| | | 5.2.8. Handling of missing data | 22 |
| 6. | PLAN | NED ANALYSIS | 23 |
| | 6.1. | STUDY POPULATION | 23 |
| | | 6.1.1. Recruited and assessable patients | 23 |
| | 6.2. | DESCRIPTION OF THE SAMPLE AT BASELINE VISIT (VISIT 1, TS) | 26 |
| | | 6.2.1. Bio-demographic characteristics | 26 |
| | | 6.2.2. Smoking history | 27 |
| | | 6.2.3. Start of COPD | 28 |
| | | 6.2.4. Exacerbations | 28 |
| | | 6.2.5. Lung function | 30 |
| | | 6.2.6. Concomitant diseases | 31 |
| | | 6.2.7. Concomitant medication | 32 |
| | | 6.2.8. Previous treatment for COPD | 33 |
| | | 6.2.9. Current treatment for COPD | 34 |

| | 6.3. | DESCRIPTION OF THE SAMPLE AFTER 6 WEEKS (VISIT 2, TS) | 35 |
|----|-------|-------------------------------------------------------|----|
| | | 6.3.1. Data after 6 weeks | 35 |
| | | 6.3.2. Treatment for COPD | 36 |
| | | 6.3.3. Concomitant diseases | 36 |
| | | 6.3.4. Concomitant medication | 37 |
| | | 6.3.5. Tobacco consumption | 38 |
| | 6.4. | ANALYSIS OF EFFICACY (FAS) | 39 |
| | | 6.4.1. Analysis of primary endpoint | 39 |
| | | 6.4.2. Analysis of secondary endpoints | 39 |
| | 6.5. | SAFETY ANALYSIS (TS) | 43 |
| | | 6.5.1. Adverse events | 43 |
| | | 6.5.2. Drug-related adverse events | 44 |
| | | 6.5.3. Serious Adverse Events | 45 |
| | | 6.5.4. Pregnancy | 46 |
| 7. | REFER | RENCES | 54 |
| 3. | ANNE | EX | 55 |
| | 8.1. | ANNEX 1. DB DEBUGGING | 55 |
| | 8.2. | ANNEX 2. DETAILS OF THE NON-ASSESSABLE PATIENTS | 56 |
| | 8.3. | ANNEX 3. RECORDED CONCOMITANT DISEASES | 57 |
| | 8.4. | ANNEX 4. CONCOMITANT MEDICATION | 62 |
| | 8.5. | ANNEX 5. PREVIOUS TREATMENT FOR COPD | 65 |
| | 8.6. | ANNEX 6. CURRENT TREATMENT FOR COPD | 67 |

# **LIST OF FIGURES**

| FIGURE 1. | GOLD VERSION 2014 | 19 |
|---|---|---|
| FIGURE 2. | GOLD VERSION 2017 | 20 |
| FIGURE 3. | FLOW CHART OF PATIENTS RECRUITED ONTO THE STUDY | 25 |
| FIGURE 4. | THERAPEUTIC SUCCESS AFTER 6 WEEKS (VISIT 2) — FULL ANALYSIS SET (FAS) | 39 |
| FIGURE 5. | PF-10 Score – Full Analysis Set (FAS) | 40 |
| FIGURE 6. | PF-10 score according to therapeutic success – Full Analysis Set (FAS) | 40 |
| FIGURE 7. | PATIENT'S GENERAL CONDITION —PGE SCORE AS ASSESSED BY THE PHYSICIAN — FULL ANALYSIS SET (FAS) | 41 |
| FIGURE 8 | PATIENT SATISFACTION WITH SPIOLTO® RESPINAT® - FULL ANALYSIS SET (FAS) | 42 |

# **LIST OF TABLES**

| TABLE 1. | IMPORTANT PROTOCOL VIOLATIONS-ALL SCREENED PATIENTS | 23 |
|---|---|---|
| TABLE 2. | INCLUSION AND EXCLUSION CRITERIA-ALL SCREENED PATIENTS | 23 |
| TABLE 3. | DISPOSITION OF PATIENTS-ALL SCREENED PATIENTS | 24 |
| TABLE 4. | ASSESSABLE PATIENTS BY VISIT AND SAMPLE SET | 24 |
| TABLE 5. | SUMMARY OF ANALYSIS POPULATION AND ENDPOINTS | 25 |
| TABLE 6. | SOCIO-DEMOGRAPHIC DATA - TREATED SET (TS) | 26 |
| TABLE 7. | Anthropometric data - Treated Set (TS) | 26 |
| TABLE 8. | Smoking history - Treated Set (TS) | 27 |
| TABLE 9. | MEDICAL HISTORY - TREATED SET (TS) | 28 |
| TABLE 10. | EXACERBATIONS IN THE LAST 12 MONTHS - TREATED SET (TS) | 28 |
| TABLE 11. | BASELINE LUNG FUNCTION (VISIT 1) - TREATED SET (TS) | 30 |
| TABLE 12. | CONCOMITANT DISEASES AT BASELINE VISIT (VISIT 1) - TREATED SET (TS) | 32 |
| TABLE 13. | CONCOMITANT MEDICATION AT BASELINE VISIT (VISIT 1) - TREATED SET (TS) | 32 |
| TABLE 14. | TREATMENT FOR COPD IN THE 6 MONTHS PRIOR TO THE BASELINE VISIT (VISIT 1) - TREATED SET (TS) | 33 |
| TABLE 15. | CURRENT TREATMENT FOR COPD - TREATED SET (TS) | 34 |
| TABLE 16. | CONTINUATION OF THE PATIENT IN THE STUDY AFTER 6 WEEKS (VISIT 2) - TREATED SET (TS) | 35 |
| TABLE 17. | CONTINUATION OF TREATMENT WITH SPIOLTO® RESPIMAT® AFTER 6 WEEKS (VISIT 2) - TREATED SET (TS) | 36 |
| TABLE 18. | NEW CONCOMITANT DISEASES AFTER 6 WEEKS (VISIT 2) - TREATED SET (TS) | 36 |
| TABLE 19. | Additional concomitant medication after 6 weeks (visit 2) - Treated Set (TS) | 37 |
| TABLE 20. | Tobacco consumption after 6 weeks (visit 2) - Treated Set (TS) | 38 |
| TABLE 21. | THERAPEUTIC SUCCESS AFTER 6 WEEKS (VISIT 2) — FULL ANALYSIS SET (FAS) | 39 |
| TABLE 22. | PF-10 SCORE AT BASELINE VISIT, AFTER 6 WEEKS AND CHANGE – FULL ANALYSIS SET (FAS) | 39 |
| TABLE 23. | CHANGE IN PF-10 SCORE ACCORDING TO THERAPEUTIC SUCCESS – FULL ANALYSIS SET (FAS) | 40 |
| TABLE 24. | GENERAL CONDITION OF THE PATIENT – PGE SCORE AS ASSESSED BY THE PHYSICIAN AT THE BASELINE VISIT AND A | FTER |
| | 6 WEEKS IN COMPLETED PATIENTS — FULL ANALYSIS SET (FAS) | 40 |
| TABLE 25. | PATIENT SATISFACTION WITH SPIOLTO® RESPIMAT® AFTER 6 WEEKS OF TREATMENT (VISIT 2) IN COMPLETED PATI | ENTS |
| | - FULL ANALYSIS SET (FAS) | 41 |
| TABLE 26. | ADVERSE EVENTS (AE) OVERALL SUMMARY - TREATED SET (TS) | 43 |
| TABLE 27. | AE ACCORDING TO MEDDRA-SOC AND PT - TREATED SET (TS) | 43 |
| TABLE 28. | SUMMARY DRUG-RELATED ADVERSE EVENTS - TREATED SET (TS) | 44 |
| TABLE 29. | SERIOUS DRUG-RELATED ADVERSE EVENTS - TREATED SET (TS) | 44 |
| TABLE 30. | Non-Serious Drug-related adverse events - Treated Set (TS) | 44 |
| TABLE 31. | OUTCOME DRUG-RELATED ADVERSE EVENTS - TREATED SET (TS) | 45 |
| TABLE 32. | CHARACTERISTICS OF SERIOUS ADVERSE EVENTS - TREATED SET (TS) | 45 |
| TABLE 33. | PATIENT PREGNANT AT AE - TREATED SET (TS) | 46 |


| I ABLE 48. | VALIDATION DURING DATA ENTRY: SELECTION CRITERIA | .55 |
|---|---|---|
| TABLE 49. | DEBUGGING PERFORMED DURING THE STATISTICAL ANALYSIS | .55 |
| TABLE 50. | New variables created for the preparation of the results report | .55 |
| TABLE 51. | DESCRIPTION OF THE TS NON-ASSESSABLE PATIENTS | .56 |
| TABLE 52. | DESCRIPTION OF THE FAS NON-ASSESSABLE PATIENTS | .56 |
| TABLE 53. | CONCOMITANT DISEASES AT BASELINE VISIT (VISIT 1) — TREATED SET (TS) | .57 |
| TABLE 54. | DURATION OF CONCOMITANT DISEASES AT BASELINE VISIT (MONTHS) ) — TREATED SET (TS) | .58 |
| TABLE 55. | NEW CONCOMITANT DISEASES AFTER 6 WEEKS (VISIT 2) ) — TREATED SET (TS) | .59 |
| TABLE 56. | Duration of New Concomitant diseases after 6 weeks (months) – Treated Set (TS) | .60 |
| TABLE 57. | CONCOMITANT MEDICATION AT BASELINE VISIT (VISIT 1) — TREATED SET (TS) | .62 |
| TABLE 58. | DURATION OF CONCOMITANT MEDICATION AT BASELINE VISIT (MONTHS) — TREATED SET (TS) | .62 |

| TABLE 59. | ADDITIONAL CONCOMITANT MEDICATION AFTER 6 WEEKS (VISIT 2) – TREATED SET (TS) |
|---|---|
| TABLE 60. | Duration (months) of the additional concomitant medication after 6 weeks (visit 2) — Treated Set |
| | (TS)63 |
| TABLE 61. | TREATMENT FOR COPD IN THE 6 MONTHS PRIOR TO THE BASELINE VISIT (VISIT 1) - ACTIVE SUBSTANCE — TREATED |
| | SET (TS) |
| TABLE 62. | DURATION OF TREATMENT FOR COPD IN THE 6 MONTHS PRIOR TO THE BASELINE VISIT (VISIT 1) - ACTIVE SUBSTANCE |
| | - Treated Set (TS)66 |
| TABLE 63. | CURRENT TREATMENT FOR COPD (VISIT 1) — TREATED SET (TS) |
| TABLE 64. | CURRENT TREATMENT FOR COPD (VISIT 2) — TREATED SET (TS) |
| TABLE 65. | Individualised description of the adverse events under study — Treated Set (TS) |
| TABLE 66. | Individualised description of the serious adverse events under study – Treated Set (TS) |

## 2. GLOSSARY OF ABBREVIATIONS

The meanings of the abbreviations used in this document are explained below:

**95% CI** 95% confidence interval

AE Adverse event

AR Adverse reaction to the drug

**COPD** Chronic obstructive pulmonary disease

**CRA** Clinical Research Associate

**CRF** Case report form

DMP Data management plan
eCRF Electronic case report form

**FEV1** Forced expiratory volume in one second

GOLD Global Initiative for Chronic Obstructive Lung Disease

ICH International Conference on Harmonisation

ICF Informed consent form
ICS Inhaled corticosteroids

IEC Independent Ethics Committee

LABA Long-acting beta<sub>2</sub> adrenoceptor agonist
LAMA Long-acting muscarinic antagonist

**LCM** Local Clinical Monitor

Max Maximum

MedDRA Medical Dictionary for Regulatory Activities

Min Minimum

mMRC Modified Medical Research Council Scale

**p** p-value associated with the statistical test used

P25-P75 25th percentile - 75th percentile
PASS Power Analysis & Sample Size

**PF-10** Physical Functioning patient questionnaire

PGE Physician's Global Evaluation

**SAE** Serious adverse event

SAMA Short-acting muscarinic antagonist

SAP Statistical Analysis Plan
SAS Statistical Analysis System

SD Standard deviation

**SF-36** 36-Item Short Form Health Survey

Date: 18/02/2019 (Final Version 2.0) CONFIDENTIAL Página 12 de 68

## 3. STUDY OBJECTIVES

## **3.1.** PRIMARY OBJECTIVE

The primary objective of the study is to measure changes in physical functioning - serving as a surrogate for physical activity and exercise capacity - in COPD patients being treated with Spiolto® Respimat® after approximately 6 weeks.

## 3.2. SECONDARY OBJECTIVES

The secondary objectives are to assess the changes in PF-10 score from visit 1 (baseline visit at start of the study) to visit 2 (final visit, approximately 6 weeks after visit 1), the patient's general condition (physician's assessment – PGE score) at visit 1 and at visit 2, as well as patient satisfaction with Spiolto® Respimat® at visit 2.

Date: 18/02/2019 (Final Version 2.0) CONFIDENTIAL Página 13 de 68

4. STUDY POPULATION

It is expected that data will be collected from approximately 1000 patients at approximately 200 sites

(primary care centres) in Spain. Sites will be selected in a way that reflects routine clinical practice for

COPD in order to ensure the representativeness of the population with COPD. The inclusion of 5

patients per investigator has been planned.

A record will be kept of all patients included in the study (i.e., who have given their informed consent)

in the investigating site's file, irrespective of whether they have been treated or not.

4.1. SELECTION CRITERIA

Patients who meet all the criteria listed below may be included:

4.1.1. Inclusion criteria

1. Written informed consent prior to participation

2. Female and male patients ≥ 40 years of age

3. Patients diagnosed with COPD and requiring long-acting dual bronchodilation

(LAMA + LABA) treatment according to approved Spiolto® Respimat® SmPC and

COPD GOLD guideline recommendation

4.1.2. Exclusion criteria

1. Patients with contraindications according to Spiolto® Respimat® SmPC

2. Patients who have been treated with a LABA/LAMA combination (free and fixed

dose) in the previous 6 months

3. Patients continuing LABA-iCS treatment should not be additionally treated with

Spiolto® Respimat® in order to avoid a double dosing of long-acting beta-agonists

4. Patients for whom further follow-up is not possible at the enrolling site during the

planned study period of approx. 6 weeks

5. Pregnancy and lactation

6. Patients currently listed for lung transplantation

7. Current participation in any clinical trial or any other non-interventional study of a

drug or device

4.2. RATIONALE FOR SAMPLE SIZE

In a previous study, 205.426 (clinicaltrials.gov NCT 00699699: "Assessment of Physical Activity

(PF10 Sub Domain of SF-36 Activity Score) and Tolerability in COPD Patients During Treatment

With Spiriva® Respimat®)", with more than 1000 patients treated with Spiriva® Respimat®,

therapeutic success (i.e., 10-point increase in the PF-10 score between visit 1 and visit 2) was

achieved in 61% of patients.

In this study, a lower therapeutic success rate is expected, as patients may already be on

maintenance treatment at the start. Assuming a therapeutic success rate of 50% and 900

patients, the 95% confidence interval for the therapeutic success rate would be between 46.7%

(lower limit) and 53.3% (upper limit) (level of accuracy of ± 3.3%), basing the calculations on a

normal approximation to the binomial distribution.

Taking into account a possible drop-out rate of 10%, the sample size is adjusted to 1000

patients.

Calculations were made using the PASS software package, version 2011.

OTIVACTO (1237.58) - SAP

Date: 18/02/2019 (Final Version 2.0) CONFIDENTIAL Página 15 de 68

## 5. METHODS

# **5.1.** DATA PROCESSING

The data management process detailed in the Data Management Plan (DMP) for studies conducted only in electronic format, includes the coding and the definition of the filters for the validation of data during the tabulation of the data or once in tabulated form.

## **5.2.** DATA ANALYSIS AND STATISTICAL TESTS

## **5.2.1.** Important protocol violations

The next table defines the different categories of important protocol violations (PVs). The final column describes which PVs will be used to exclude subjects from the different patient analysis sets:

| Description | Requirements | Excluded from |
|---|---|---|
| Entrance criteria not met | | |
| Inclusion criterion 1 (Written informed consent prior to participation) | not met as specified in the protocol | None |
| Inclusion criterion 2 (Female and male patients ≥ 40 years of age) | not met as specified in the protocol | None |
| Inclusion criterion 3 (Patients diagnosed with COPD and requiring long-<br>acting dual bronchodilation (LAMA + LABA) treatment according to<br>approved Spiolto® Respimat® SmPC and COPD GOLD guideline<br>recommendation) | not met as specified in the protocol | None |
| Exclusion criterion 1 (Patients with contraindications according to Spiolto® Respimat® SmPC) | met as specified in the protocol | None |
| Exclusion criterion 2 (Patients who have been treated with a LABA/LAMA combination (free and fixed dose) in the previous 6 months) | met as specified in the protocol | None |
| Exclusion criterion 3 (Patients continuing LABA-ICS treatment should not be additionally treated with Spiolto® Respimat® in order to avoid a double dosing of long-acting beta-agonists) | met as specified in the protocol | None |
| Exclusion criterion 4 (Patients for whom further follow-up is not possible at the enrolling site during the planned study period of approx. 6 weeks) | met as specified in the protocol | None |
| Exclusion criterion 5 (Pregnancy and lactation) | met as specified in the protocol | None |
| Exclusion criterion 6 (Patients currently listed for lung transplantation) | met as specified in the protocol | None |
| Exclusion criterion 7 (Current participation in any clinical trial or any other non-interventional study of a drug or device) | met as specified in the protocol | None |
| Informed consent | | |
| Informed consent not available/not done | Inclusion criterion not met as specified in the protocol or informed consent date missing | All |

**5.2.2.** Population for analysis

Three populations will be used for the analysis:

1. All screened patients: defined as all recruited patients with informed consent and date of

registration.

2. Treated Set (TS): All screened patients with at least one documented administration of

Spiolto Respimat. This population will be used in the safety endpoints,

demographics/baseline, and other summary tables.

3. Full Analysis Set (FAS): All screened patients with at least one documented administration

of Spiolto Respimat and available PF-10 score at visit 1 and visit 2. This population will be

used in the primary and secondary tables,

5.2.3. Analysis of primary endpoint

For the primary endpoint, the proportion of patients with therapeutic success at visit 2 i.e.,

approximately 6 weeks (define as 10-point increase in the PF-10 score between visit 1 and visit

2) together with the 95% confidence interval will be presented.

\***PF-10** is a sub-domain of SF-36 and consists of 10 items evaluating the scope of the restrictions

experienced when carrying out routine activities. Each PF-10 item may be answered with "yes,

limited a lot", "yes, limited a little", or "no, not limited at all", with a score of 1, 2 or 3. The

scores of the 10 items are added up, resulting in a value between 10 (a patient who answers

all questions with "yes, limited a lot") and 30 (a patient who answers all questions with "no,

not limited at all"). The final sum of the individual scores will be standardised to a range of 0 to

100 using the following formula: 100x(sum-10)/20.1

5.2.4. Analysis of secondary endpoints

The secondary endpoints are listed below:

Changes in PF-10 score from visit 1 to visit 2

- Patient's general condition assessed by the physician (PGE score) at visit 1 and visit 2.

- Patient satisfaction with Spiolto® Respimat® at visit 2.

The head physician will use the Physician's Global Evaluation (PGE) to assess the patient's

general condition on an 8-point ordinal scale from 1 (very poor) to 8 (excellent). The PGE will

be completed before and approximately 6 weeks after the start of treatment.

A patient satisfaction questionnaire will also be completed during visit 2, using a 7-point

ordinal scale, from 1 (very unsatisfied) to 7 (very satisfied).

5.2.5. Analysis of other endpoints

In addition, at visit 1 and/or visit 2 the following parameters will be analysed:

• Patient demographic data (age, gender, height and weight)

Smoking history

• Reported exacerbations

Dyspnoea based on the mMRC score at visit 1

• GOLD spirometric classification (1, 2, 3, 4)

• GOLD group of patients (A, B, C, D)

Comorbidities

Medication related to COPD and other concomitant medication

• Details of treatment with inhaled drugs for the airways prior to the study

Details of treatment with inhaled drugs for the airways during the study

• Reasons for ending treatment during the observation period

• Details of treatment continuation/discontinuation

Adverse reactions to the drug (AR and SAR), fatal AEs, pregnancies

Medical history collected during routine clinical care will be used to evaluate patient

inclusion/exclusion criteria. These medical histories will be used to collect patient demographic

data, smoking history, prior medications for COPD, concomitant diseases and concomitant

medication.

The mMRC scale will be used to assess the status of the patient's dyspnoea before and after

treatment.

GOLD group (A, B, C, D) of patients will be analyzed according:

GOLD version 2014 – COPD degree of severity (GOLD group)<sup>2</sup>:

As detailed above, the CAT is recommended as a comprehensive measure of symptoms, with

a CAT score ≥ 10 indicating a high level of symptoms. Comprehensive assessment of the

symptomatic impact of the disease is preferred, but in its absence mMRC scores provide an assessment of the impact of dyspnoea. It is unnecessary and possible confusing to use more than one scale.

There are three methods of assessing exacerbation risk. <u>One</u> is the population-base method using the GOLD spirometric classification, with GOLD 3 or GOLD 4 categories indicating high risk. The <u>second</u> based on the individual patient's history of exacerbations, with two or more exacerbations in the preceding year indicating high risk. The <u>third</u> is a history of hospitalization due to an exacerbation in the preceding year. If there is a discrepancy between these criteria, the assessment pointing to the highest risk should be used.



Figure 1. GOLD version 2014

2. GOLD version 2017 – COPD degree of severity (GOLD group)<sup>3</sup>- Based on symptoms and exacerbations only

A refinement of the ABCD assessment tool is proposed in the 2017 GOLD Report that separates spirometric grades from the ABCD groups. ABCD groups and their associated for pharmacotherapy recommendations will be derived exclusively from patients symptoms and their history of exacerbations.

In the refined assessment scheme, patients should undergo spirometry to determine the severity of airflow limitations (i.e. spirometric grade). They should also undergo assessment of their dyspnoea using mMRC or symptoms using CAT. Finally, their history of exacerbations

(including prior hospitalizations) should be recorded. The number provides information regarding severity of airflow limitation (spirometric grade 1 to 4) while the letter (groups A to D) provides information regarding symptom burden and the risk of exacerbation which can be used to guide therapy.

Figure 2. GOLD version 2017



5.2.7. Statistical methodology

In this observational study, cross-sectional data will be collected at the start of the study and

longitudinal follow-up data will be collected in the 6-week period for patients with COPD

disease requiring dual bronchodilator therapy in routine clinical practice.

Baseline data will be described using a cross-sectional approach. Longitudinal follow-up data

will be summarised descriptively. Due to the observational nature of this study, it is not planned

to carry out (confirmatory) hypothesis testing in a strict statistical sense. Analyses are

descriptive in nature and confidence intervals and p-values from statistical models will be used

for exploratory purposes. No adjustments for multiple testing will be carried out in the

statistical significance evaluation. Consequently, significant differences may be observed by

chance along and p-values should be interpreted as exploratory and treated with caution. No

formal hypothesis testing will be performed as this is a self-controlled study.

The statistical characteristics presented in the results tables will include: N (total number of

valid values), mean, standard deviation (SD), 95% confidence interval of the mean (95% CI),

median, 25th and 75th percentiles (P25 and P75, respectively), minimum and maximum (min

and max, respectively) for continuous endpoints. The categorical endpoints will be described

by their absolute and relative frequencies. The proportion rates and the 95%CIs will be

provided when appropriate.

For the primary endpoint, the proportion of patients with therapeutic success at visit 2 (a 10-

point increase in the PF-10 score between visit 1 and visit 2) together with the 95% confidence

interval will be presented.

For the secondary endpoints:

Changes in PF-10 score from visit 1 to visit 2

- Patient's general condition assessed by the physician (PGE score) at visit 1 and visit 2.

Patient satisfaction with Spiolto® Respimat® at visit 2.

The patient's general condition (PGE score) at visit 1 and visit 2, the mMRC at visit 1 and patient

satisfaction at visit 2 are categorical endpoints, so they will be analysed in frequency tables.

The change from visit 1 to visit 2 in the PF-10 score is a continuous assessment criterion, so it

will be analysed by: n (total number of valid values), mean, standard deviation (SD), 95%

confidence interval of the mean (95% CI), median, 25th and 75th percentiles (P25 and P75,

respectively), minimum and maximum (min and max, respectively).

Changes in the PF-10 between visit 1 and visit 2 will be analysed using a paired t-test or the

non-parametric Wilcoxon Rank-Sum Test for data with non-normal distribution). Changes in

the PGE between visit 1 and visit 2 will be analysed using McNemar test.

Data on safety will be reported according to local requirements. Statistical analyses and

reporting of adverse reactions (ARs)/adverse events (AEs) will be descriptive in nature. The

incidences of ARs and AEs will be analysed in relation to the number of treated patients.

Every effort will be made to collect complete data at the specified study visits (see DMP). Any

data removed from the analysis will be documented, recording the site and the patient

number, as well as the reason for the removal (see the ANNEX 1. DB DEBUGGING).

A statistical significance level of 0.05 will be applied in all the statistical tests. The evaluation

will be carried out using SAS® software, version 9.4 or later.

5.2.8. Handling of missing data

In context of PF-10 questionnaire, if less than half of the items on the PF-10 for a patient are

missing, the missing values will be replaced with the mean of the other values and the PF-10

score will be calculated. If half or more of the items on the PF-10 are missing, no score will be

calculated and the PF-10 score will be marked as not available.

No other missing data will be imputed. If patients have missing values for any other endpoints,

these patients will be excluded from the analysis of that endpoint.

## **6.1. STUDY POPULATION**

## 6.1.1. Recruited and assessable patients

According to the section 5.2.2, three populations will be used for the analysis: All screened patients, Treated Set (TS) and Full Analysis Set (FAS). Details of patients excluded from the TS and patients excluded from the FAS will be included in Annex 2, section 8.2.

The important protocol violations will be described in the following table:

| Table 1. | Important protocol violations-All screened patients | | |
|---|---|---|---|
| | | n | % |
| Total patients | | | 100.0 |
| | of informed consent (IC-1) | | |
| Total with violation | of any other inclusion criterion | | |
| Total with violation | of any exclusion criterion | | |
| Total with violation | of any inclusion or exclusion criterion | | |

The inclusion criteria and exclusion criteria based on all screened patients according to CRFs:

| Table 2. | Inclusion and Exclusion criteria-A | All screened pati | ents | |
|---|---|---|---|---|
| | | | n | % |
| Total patients at screen | | | | |
| Inclusion criteria not fulfilled | | | | |
| IC1. Written informed consen | t prior to participation | | | |
| IC2. Female and male patient | s ≥ 40 years of age | | | |
| _ | COPD and requiring dual bronchodil<br>ording to approved Spiolto® Respinendation | | | |
| <b>Exclusion criteria fulfilled</b> | | | | |
| EC1. Patients with contraindic | ations according to Spiolto® Respin | nat® SmPC | | |
| EC2. Patients who have been and fixed dose) in the previou | treated with a LABA/LAMA combina<br>s 6 months | ation (free | | |
| _ | /ICS treatment should not be addit<br>at® in order to avoid a double dosin | • | | |
| EC4. Patients for whom furthed during the planned study perior | er follow-up is not possible at the er<br>od of approx. 6 weeks | nrolling site | | |
| EC5. Pregnancy and lactation | | | | |
| EC6. Patients currently listing | for lung transplantation | | | |

| Table 2. | Inclusion and Exclusion criteria-All scr | eened patients | |
|---|---|---|---|
| | | n | % |
| EC7. Current participation in interventional study of a dru | n any clinical trial or any other non-<br>ug or device | | |

The disposition of patient will be described in the following table:

| Table 3. | Disposition of patients-All scr | eened patie | nts |
|---|---|---|---|
| | | n | % |
| Total patients at screen | | | |
| Total patients at visit 1 | | | |
| Total patients at visit 2 | | | |
| <b>Total patients on Reaso</b> | n for not performing visit 2 | | |
| Adverse event | | | |
| Serious adverse even | t | | |
| Patient's wish | | | |
| Withdrawn consent | | | |
| Lost to follow-up | | | |
| Patient died | | | |
| Other | | | |
| Total patients for discor | ntinuation | | |
| Lost to follow-up | | | |
| Not meet inclusion/ex | xclusion criteria | | |
| Adverse event | | | |
| Protocol deviation | | | |
| Patient's wish | | | |
| Investigator's wish | | | |
| Other | | | |

The following table describes the number of assessable patients with data in visit 1 and visit 2 according the sample sets (screened patients, TS, FAS):

| | Table 4. | Assessable patients by visit and sample set | | |
|---|---|---|---|---|
| | Recruited<br>patients<br>n (%) | All screened<br>patients<br>n (%) | Assessable patients in TS n (%) | Assessable patients<br>in FAS<br>n (%) |
| Visit 1 | | | | |
| Visit 2 | | | | |

All screened patients: All recruited patients with informed consent and date of registration.

 $\label{thm:condition} \textbf{Treated Set (TS): All screened patients with at least one documented administration of Spiolto^{@}\ Respirat^{@}.}$ 

Full Analysis Set (FAS): All screened patients with at least one documented administration of Spiolto® Respimat® and available PF-10 score at visit 1 and visit 2.



Figure 3. Flow chart of patients recruited onto the study

\*In context of PF-10 questionnaire, if less than half of the items on the PF-10 for a patient are missing, the missing values will be replaced with the mean of the other values and the PF-10 score will be calculated. If half or more of the items on the PF-10 are missing, no score will be calculated and the PF-10 score will be marked as not available.

In the ANNEX 2. DETAILS OF THE NON-ASSESSABLE PATIENTS, the lists of the non-assessable patients in TS and FAS will be specified.

| | Table | 5. | Summary of analysis population and endpoints | | | | |
|---|---|---|---|---|---|---|---|
| | n | % | Baseline characteristics | Characteristics after 6 weeks | Primary endpoint | Secondary endpoints | Safety<br>endpoints |
| Treated Set (TS) | | | X | Х | | | Х |
| Full Analysis Set (FAS) | | | | | Х | Х | |

All screened patients: All recruited patients with informed consent and date of registration.

Treated Set (TS): All screened patients with at least one documented administration of Spiolto® Respimat®.

Full Analysis Set (FAS): All screened patients with at least one documented administration of Spiolto® Respimat® and available PF-10 score at visit 1 and visit 2.

# **6.2.** DESCRIPTION OF THE SAMPLE AT BASELINE VISIT (VISIT 1, TS)

This section will describe the socio-demographic characteristics, anthropometric data, smoking history and baseline characteristics in terms of the COPD diagnosis, exacerbations, lung function, concomitant diseases, concomitant medication, and previous and current treatment for COPD of the **Treated Set (TS)** (n=xxx) (see Table 4).

#### **6.2.1.** Bio-demographic characteristics

This section will describe the socio-demographic data and anthropometric data of the treated patients being studied.

| Table 6. | Socio-demographic data - Treated Set (TS) |
|-------------------------|-------------------------------------------|
| | Total |
| Age (years) | |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |
| Pooled age n (%) | |
| < 65 years | |
| ≥ 65 years | |
| Gender n (%) | |
| Male | |
| Female | |
| Employment status n (%) | |
| Working | |
| Unemployed | |
| Temporarily unable to w | rork |
| Permanently unable to v | vork |
| Retired | |
| Other <sup>1</sup> | |

<sup>&</sup>lt;sup>1</sup>Specify 'other':

| | | Table | 7. | Anthropo | metric data - Treated S | et (TS) | | |
|---|---|---|---|---|---|---|---|---|
| | n | mean | SD | (95% CI) | Median [P25; P75] | Min | Max | p¹ |
| Weight (kg) | | | | | | | | |
| Male | | | | | | | | |
| Female | | | | | | | | |
| Height (cm) | | | | | | | | |
| Male | | | | | | | | |
| Female | | | | | | | | |
| BMI (kg/m²) | | | | | | | | |

| | | Table 7. | | Anthropometric data - Treated Set (TS) | | | | |
|---|---|---|---|---|---|---|---|---|
| | n | mean | SD | (95% CI) | Median [P25; P75] | Min | Max | p <sup>1</sup> |
| Male | | | | | | | | |
| Female | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Student's t-test/Mann-Whitney U test

## 6.2.2. Smoking history

This section will describe the smoking history of the assessable patients being studied.

| | Table 8. | Smoking history - Treated Set (TS) |
|----------------|---------------------|------------------------------------|
| | | Total |
| Smoking n (%) | | |
| Non-smoker | | |
| Ex-smoker | | |
| Smoker | | |
| Number of pack | -years - Ex-sm | oker |
| Mean (SD) | | |
| 95% CI | | |
| Median (P25; P | 75) | |
| (Min; Max) | | |
| N | | |
| Number of pack | -years - Smok | er |
| Mean (SD) | | |
| 95% CI | | |
| Median (P25; P | 75) | |
| (Min; Max) | | |
| N | | |
| Number of pack | -years <sup>1</sup> | |
| Mean (SD) | | |
| 95% CI | | |
| Median (P25; P | 75) | |
| (Min; Max) | | |
| N | | |

<sup>&</sup>lt;sup>1</sup> Sample of ex-smokers and smokers (n=xx)

Pack-years = (number of cigarettes smoked per day x number of smoking years) / 20

#### 6.2.3. Start of COPD

This section will describe the time from the diagnosis of COPD to the baseline visit (visit 1).

| Table 9. | Medical history - Treated Set (TS) |
|-----------------------------|------------------------------------|
| | Total |
| Time from COPD diagnosis to | date of baseline visit |
| (years) | |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |

## 6.2.4. Exacerbations

This section will describe the exacerbation episodes, attendance at the emergency department and hospital admission which have occurred in the last 12 months relative to the baseline visit (visit 1).

| Table 10. | Exacerbations in the last 12 months - Treated Set (TS) |
|---|---|
| | Total |
| · | nced any moderate COPD<br>nich required corticosteroids<br>s)? n (%) |
| Yes | |
| No | |
| Unknown | |
| Number of moderate exace | erbation episodes <sup>1</sup> |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |
| Frequency of moderate exa | acerbation episodes <sup>1</sup> n (%) |
| 0 | |
| 1 | |
| 2 | |
| Function and a section and a s | and the state of t |
| Frequency of moderate exa<br>≤ 1 exacerbation episode | acerbation episodes n (%) |
| ≥ 2 exacerbation episodes | |
| Time from the last episode | |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N N | |

| Table 10. | Exacerbations in the last 12 months - Treated Set (TS) |
|---|---|
| | Total |
| | the emergency department |
| because of COPD (exacer | bation)? n (%) |
| Yes | |
| No | |
| Unknown | |
| He/she came to the en<br>Primary setting <sup>2</sup> n (%) | nergency department in the |
| | nergency department in the |
| Hospital setting <sup>2</sup> n (%) | |
| | ne came to the emergency |
| department in the Primar<br>Mean (SD) | y setting |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max)<br>N | |
| | to the emergence |
| department in the Hospit | ne came to the emergency |
| Mean (SD) | ai setting |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max)<br>N | |
| | witel administra because of |
| his/her COPD (severe exa | spital admission because of |
| Yes | cerbaneny: II (70) |
| No | |
| Unknown | |
| Number of hospitalisation | ns that he/she has had <sup>5</sup> |
| Mean (SD) | is that he/she has had |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |
| Total number of days adn | nitted <sup>5</sup> |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |
| Time from the last hospit | alisation until visit 1 |
| (months) <sup>5</sup> | ANDALISH WHEN VISIC I |
| Mean (SD) | |

| Table 10. | Exacerbations in the last 12 months - Treated Set (TS) |
|-------------------|--------------------------------------------------------|
| | Total |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |

<sup>&</sup>lt;sup>1</sup> If the patient has experienced any moderate exacerbation episodes (n=xx)

## 6.2.5. Lung function

This section will describe the lung function of the patient at the baseline visit (visit 1).

| Table 11. | Baseline lung function (visit 1) - Treated Set (TS) |
|---|---|
| | Total |
| Time from spirometry to | visit 1 (months) |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |
| FVC (ml) | |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |
| FVC (%) | |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max)<br>N | |
| FEV <sub>1</sub> (ml) | |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |
| FEV <sub>1</sub> (%) | |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |

<sup>&</sup>lt;sup>2</sup> If the patient came to the emergency department because of his/her COPD (n=xx)

<sup>&</sup>lt;sup>3</sup> If the patient came to the emergency department in the Primary setting (n=xx)

<sup>&</sup>lt;sup>4</sup> If the patient came to the emergency department in the hospital setting (n=xx)

<sup>&</sup>lt;sup>5</sup> If the patient required hospital admission because of his/her COPD (n=xx)

| Table 11. | Baseline lung function (visit 1) - Treated Set (TS) |
|---|---|
| | Total |
| (Min; Max) | |
| N | |
| FEV <sub>1</sub> /FVC | |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |
| mMRC Dyspnoea Sca | <b>le</b> n (%) |
| Grade 0 | |
| Grade I | |
| Grade II | |
| Grade III | |
| Grade IV | |
| <b>GOLD</b> classification o | f severity <sup>1</sup> n (%) |
| GOLD 1 (Mild) | |
| GOLD 2 (Moderate) | |
| GOLD 3 (Severe) | |
| GOLD 4 (Very sever | e) |
| GOLD version 2014 <sup>2</sup> | n (%) |
| GOLD A | |
| GOLD B | |
| GOLD C | |
| GOLD D | |
| GOLD version 2017 <sup>3</sup> | n (%) |
| GOLD A | |
| GOLD B | |
| GOLD C | |
| GOLD D | |
| <sup>1</sup> GOLD classification of 0 | COPD severity (based on post-bronchodilator FEV1): Mild: $FEV_1 \ge$ |

 $<sup>^1</sup>$ GOLD classification of COPD severity (based on post-bronchodilator FEV1): Mild: FEV $_1$  ≥ 80% of predicted value, Moderate: 50% ≤ FEV $_1$  < 80% of predicted value; Severe: 30% ≤ FEV $_1$  < 50% of predicted value

## 6.2.6. Concomitant diseases

This section will describe the concomitant diseases (CDs) of treated patients, and it will give details on whether they still have them on the date of the baseline visit (visit 1).

<sup>&</sup>lt;sup>2</sup> GOLD version 2014 group of patients: See 

<sup>&</sup>lt;sup>3</sup> GOLD version 2017 group of patients: See Figure 2

| Table 12. | Concomitant diseases at baseline visit (visit 1) - Treated Set (TS) | | | |
|---|---|---|---|---|
| | | Total <sup>1</sup> | Total with CDs <sup>2</sup> | Ongoing <sup>2</sup> |
| Does the patient present related concomitant disease | • | | | |
| Yes | | | | |
| No | | | | |
| Type of concomitant disease | se - Yes n (%) | | | |
| Cardiovascular disease | | | | |
| Diabetes mellitus | | | | |
| Musculoskeletal disorders | 5 | | | |
| Kidney diseases | | | | |
| Liver diseases | | | | |
| Osteoporosis | | | | |
| Gastro-oesophageal reflux | x (GOR) | | | |
| Lung cancer | | | | |
| Other <sup>3</sup> | | | | |

Note: Concomitant disease (CD). A patient could have more than one CD

In the ANNEX 3. RECORDED CONCOMITANT DISEASES, the diagnoses of the concomitant diseases, as well as their duration, will be specified.

#### 6.2.7. Concomitant medication

This section will describe the indication of concomitant medication (CM) of treated patients, as well as the active substance and whether they continue with treatment after the baseline visit (visit 1).

| Table 13. Concomitant medic | Concomitant medication at baseline visit (visit 1) - Treated Set (TS) | | |
|---|---|---|---|
| | Total <sup>1</sup> | Total with CM <sup>2</sup> | Ongoing <sup>2</sup> |
| Is the patient receiving any concomitant medication? n (%) | | | |
| Yes | | | |
| No | | | |
| Indication of the concomitant medication - | | | |
| <b>Yes</b> n (%) | | | |
| Indication 1 | | | |
| Indication 2 | | | |
| Indication 3 | | | |

Note: Concomitant medication (CM). The same patient could have more than one CM

<sup>&</sup>lt;sup>1</sup> Of the total number of treated patients (n=xx)

<sup>&</sup>lt;sup>2</sup> Of the total number of patients with CDs (n=xx)

<sup>&</sup>lt;sup>3</sup> Other: AAA (n=x); BBB (n=xx); ...

<sup>&</sup>lt;sup>1</sup>Of the total number of treated patients (n=xx)

<sup>&</sup>lt;sup>2</sup> Of the total number of patients with CM (n=xx)

| Table 13. | Concomitant medication at baseline visit (visit 1) - Treated Set (TS) | | |
|---|---|---|---|
| | Total <sup>1</sup> | Total with CM <sup>2</sup> | Ongoing <sup>2</sup> |

The medication for each of the indications, as well as its duration, will be specified in the ANNEX 4. CONCOMITANT MEDICATION.

#### 6.2.8. Previous treatment for COPD

This section will describe previous treatments for COPD in the 6 months prior to the baseline visit (visit 1).

| Table 14. Treatment for COPD in the 6 months prior to the baseline visit (visit 1) - Treated Set (TS) | | | |
|---|---|---|---|
| | Total <sup>1</sup> | Total COPD <sup>2</sup> | Ongoing <sup>2</sup> |
| Has the patient received treatment for COPD in the previous 6 months? n (%) | | | |
| Yes | | | |
| No | | | |
| SAMA | | | |
| Yes | | | |
| No | | | |
| SABA | | | |
| Yes | | | |
| No | | | |
| LAMA | | | |
| Yes | | | |
| No | | | |
| LABA | | | |
| Yes | | | |
| No | | | |
| ICS | | | |
| Yes | | | |
| No | | | |
| LAMA/LABA n (%) | | | |
| Yes | | | |
| No | | | |
| LABA/ICS n (%) | | | |
| Yes | | | |
| No | | | |
| Other <sup>3</sup> | | | |
| Yes | | | |
| No | | | |

NOTE: Patients treated with a LABA/LAMA combination (free and/or fixed combination) within the 6 previous months should not be selected for the study; the same applies to patients who continue with

# Table 14. Treatment for COPD in the 6 months prior to the baseline visit (visit 1) Treated Set (TS) Total Total COPD<sup>2</sup> Ongoing<sup>2</sup>

LABA/ICS treatment, who should not be treated in addition with Spiolto® Respimat® to prevent double-dosing of long-acting beta agonists (see section 4.1.2).

The drugs (active substance) for each one of the drug classes, as well as their duration, will be specified in the ANNEX 5. PREVIOUS TREATMENT FOR COPD.

#### 6.2.9. Current treatment for COPD

This section will describe the current treatment for COPD that the patients will receive.

| Table 15. Current treatment for COPD - Treated Set (TS) | | |
|---|---|---|
| | Total <sup>1</sup> | Total <sup>2</sup> |
| Is the patient going to be treated with Spiolto® Respimat®? n (%) | | |
| Yes | | |
| No | | |
| Has the patient been trained properly on how to use Respimat®? n (%) | | |
| Yes | | |
| No | | |
| Is the patient going to receive other inhaled treatments for COPD? n $(\%)$ | | |
| Yes | | |
| No | | |
| Other inhaled treatments for COPD¹ n (%) | | |
| SABA | | |
| ICS | | |

NOTE: All treated patients must have received a dose of the study treatment

The ANNEX 6. CURRENT TREATMENT FOR COPD will specify the concomitant medication prescribed for COPD and its duration.

<sup>&</sup>lt;sup>1</sup> Of the total number of treated patients (x = xx)

<sup>&</sup>lt;sup>2</sup> Of the total number of patients who have received treatment for COPD in the previous 6 months (n=xx)

<sup>&</sup>lt;sup>3</sup> Other: AAA (n=x); BBB (n=x); ...

<sup>&</sup>lt;sup>1</sup> Of the total number of patients (n=xxx)

<sup>&</sup>lt;sup>2</sup> If the patient has received another treatment for COPD (n=xx)

# 6.3. DESCRIPTION OF THE SAMPLE AFTER 6 WEEKS (VISIT 2, TS)

This section will describe the follow-up of patients after 6 weeks of the study and the changes which occurred after 6 weeks of treatment with Spiolto® Respimat® (treatment for COPD, concomitant diseases and medication, smoking habit, etc.) of the Treated Set (TS) and those with data at the visit after 6 weeks (see Table 4).

#### 6.3.1. Data after 6 weeks

This section will describe the number of patients who have completed their visit after 6 weeks (visit 2), the reason for discontinuation if they have not attended the visit and the time between visits (approx. 6 weeks).

| Table 16. | Continuation of the patient in the study after 6 weeks (visit 2) - Treated Set (TS) |
|---|---|
| | Total |
| Is the patient continu | ing in the study n (%) |
| Yes | |
| No | |
| Lost to follow-up | |
| Does not meet in | clusion/exclusion criteria |
| Adverse event | |
| Protocol deviation | 1 |
| Patient's decision | |
| Investigator's dec | rision |
| Other <sup>1</sup> | |
| Time between visits ( | weeks) <sup>2</sup> |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |
| Time to early termina | tion (weeks) <sup>3</sup> |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |

Specify others: other 1 (n=x); other 2 (n=x); ...

<sup>&</sup>lt;sup>2</sup> If the patient continues in the study (n=xx)

<sup>&</sup>lt;sup>3</sup> If the patient does not continue in the study (n=xx)

## 6.3.2. Treatment for COPD

This section will describe the continuity of the treatment received for COPD started at the baseline visit and the change in concomitant medication for COPD.

| Table 17. | Continuation of treatment with Spiolto<br>weeks (visit 2) - Treated Set (TS) | o® Respimat® after 6 |
|---|---|---|
| | | Total |
| | | n (%) |
| Is the patient continuing t<br>Respimat® started at the | to receive the treatment with Spiolto®<br>baseline visit? | |
| Yes | | |
| No | | |
| Reason why the patient Respimat®1 | nt is <u>no</u> longer receiving Spiolto® | |
| Reason 1 | | |
| Reason | | |
| | nedication for COPD changed with or is the patient receiving a new | |
| Yes | | |
| SABA | | |
| ICS | | |
| No | | |

<sup>&</sup>lt;sup>1</sup> If the patient is no longer receiving the treatment with Spiolto® Respimat® started at the baseline visit (n=xx)

The ANNEX 6. CURRENT TREATMENT FOR COPD 6 will specify the new concomitant medication prescribed for COPD and its duration.

## 6.3.3. Concomitant diseases

This section will describe the presence of any new concomitant diseases with respect to those of the last visit.

| Table 18. | New concomitant diseases after 6 weeks (visit 2) - Treated Set (TS) | | | |
|---|---|---|---|---|
| | | Total <sup>1</sup> | Total with new CD <sup>2</sup> | Ongoing <sup>2</sup> |
| Does the patient have a diseases with respect to t n (%) | • | | | |
| Yes<br>No | | | | |
| Table 18. New conco | New concomitant diseases after 6 weeks (visit 2) - Treated Set (TS) | | | | |
|---|---|---|---|--|--|
| | Total <sup>1</sup> | Total with<br>new CD <sup>2</sup> | Ongoing <sup>2</sup> | | |
| Type of new concomitant disease - Yes | s n (%) | | | | |
| Cardiovascular disease | | | | | |
| Diabetes mellitus | | | | | |
| Musculoskeletal disorders | | | | | |
| Kidney diseases | | | | | |
| Liver diseases | | | | | |
| Osteoporosis | | | | | |
| Gastro-oesophageal reflux (GOR) | | | | | |
| Lung cancer | | | | | |
| Other <sup>3</sup> | | | | | |

Note: Concomitant disease (CD). A patient could have more than one CD

The ANNEX 3. RECORDED CONCOMITANT DISEASES will specify the diagnoses of new concomitant diseases, as well as their duration.

#### 6.3.4. Concomitant medication

The additional intake of concomitant medication will be described in this section.

| Table 19. | Additional concomitant medication after 6 weeks (visit 2) - Treated Set (TS) | | |
|---|---|---|---|
| | Total <sup>1</sup> | Total with additional CM <sup>2</sup> | Ongoing <sup>2</sup> |
| Is the patient receiving medication? n (%) | any additional concomitant | | |
| Yes | | | |
| No | | | |
| Indication of the conco | mitant medication - Yes n | | |
| Indication 1 | | | |
| Indication 2 | | | |
| Indication 3 | | | |

Note: Concomitant medication (CM)

The additional medication for each of the indications, as well as its duration, will be specified in the ANNEX 4. CONCOMITANT MEDICATION.

<sup>&</sup>lt;sup>1</sup> Of the total number of treated patients (n=xx)

<sup>&</sup>lt;sup>2</sup> Of the total number of patients with new CD (n=xx)

<sup>&</sup>lt;sup>3</sup> Other: AAA (n=x); BBB (n=x); ...

<sup>&</sup>lt;sup>1</sup>Of the total number of treated patients (n=xx)

<sup>&</sup>lt;sup>2</sup> Of the total number of patients with additional CM (n=xx)

### 6.3.5. Tobacco consumption

This section will describe whether the patient has changed his/her smoking habits since the last visit.

| Table 20. | Tobacco consumption after 6 weeks (visit 2) - Treated Set (TS) |
|---|---|
| | Total |
| Has he/she changed his, | her smoking habits since the |
| last visit? n (%) | |
| Yes | |
| No | |
| Change of smoking habit | ¹ n (%) |
| He/she has quit smokin | g |
| He/she is smoking less | |
| He/she is smoking more | غ الماريخ الما |
| Number of cigarettes/da | y in patients who are smoking |
| less | |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |
| Number of cigarettes/da | y in patients who are smoking |
| more | |
| Mean (SD) | |
| 95% CI | |
| Median (P25; P75) | |
| (Min; Max) | |
| N | |

<sup>&</sup>lt;sup>1</sup> Of the total number of patients who have changed their smoking habit (n=xx)

Date: 18/02/2019 (Final Version 2.0) CONFIDENTIAL Página 38 de 68

 $<sup>^{2}</sup>$  Of the sample of patients who are ex-smokers and smokers in the visit after 6 weeks (n=xx). The pack-years value from the baseline visit is taken as the value in patients who have not changed their smoking habit

# 6.4. ANALYSIS OF EFFICACY (FAS)

This section will describe the results for the study's primary objective as well as for the secondary endpoints in **Full Analysis Set (FAS)**.

### 6.4.1. Analysis of primary endpoint

This section will describe the frequency and percentage of "Therapeutic success" at visit 2 (defined as: 10-point increase in the PF-10 score between the baseline visit (visit 1) and the visit after 6 weeks (visit 2) will be presented together with the 95% confidence interval.

| Table 21. | Therapeutic success after 6 weeks (visit 2) – Full Analysis Set (FAS) | |
|---|---|---|
| | Total n (%) | CI (95%) |
| Therapeutic success <sup>1</sup> n | (%) | |
| Therapeutically succe | ssful | |
| Not therapeutically su | uccessful | |

Therapeutic success: 10-point increase in the PF-10 score between visit 1 and visit 2.

Figure 4. Therapeutic success after 6 weeks (visit 2) – Full Analysis Set (FAS) [pie chart]

### 6.4.2. Analysis of secondary endpoints

This section will describe the data corresponding to the secondary efficacy endpoints.

### Changes in PF-10 score

A descriptive analysis of the PF-10 score from the baseline visit (visit 1) to the visit after 6 weeks (visit 2), as well as the change (difference visit 2 - visit 1), will be conducted in this section.

| | Table 22. | PF | -10 score at | baseline | visit, after | 6 weeks an | ıd change – Fu | II Analysi | s Set (FAS | ) |
|---|---|---|---|---|---|---|---|---|---|---|
| | | n | mean | SD | (95% CI) | Median | [P25-P75] | Min | Max | $P^1$ |
| Baseline<br>(Visit 1)<br>PF-10 aft<br>weeks (Visit | | | | | | | | | | - |
| Change in (v2-v1) | PF-10 | | | | | | | | | |

 $<sup>^{\</sup>it 1}$  paired t-test /Wilcoxon Rank-Sum

OTIVACTO (1237.58) - SAP

<sup>&</sup>lt;sup>1</sup> Of the total number of patients who have PF-10 data at the baseline visit (visit 1) and at the visit after 6 weeks (visit 2)

### Figure 5. PF-10 Score – Full Analysis Set (FAS)

[line/bar charts of the mean/median PF-10 at the baseline visit (visit 1) and the visit after 6 weeks (visit 2)]

| Table 23. | Chan | ge in PF-1 | LO scor | e according | to therape | utic success - | - Full An | alysis Set ( | (FAS) |
|---|---|---|---|---|---|---|---|---|---|
| | n | mean | SD | (95% CI) | Median | [P25-P75] | Min | Max | $P^1$ |
| Baseline PF-10 (visit 1) | | | | | | | | | |
| Therapeutically | | | | | | | | | |
| successful | | | | | | | | | |
| Not therapeutically | | | | | | | | | |
| successful | | | | | | | | | |
| PF-10 after 6 weeks | | | | | | | | | |
| (visit 2) | | | | | | | | | |
| Therapeutically | | | | | | | | | |
| successful | | | | | | | | | |
| Not therapeutically | | | | | | | | | |
| successful | | | | | | | | | |
| Change in PF-10 (v2-v1) | | | | | | | | | |
| Therapeutically | | | | | | | | | |
| successful | | | | | | | | | |
| Not therapeutically | | | | | | | | | |
| successful | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> independent two-sample t-test/Mann–Whitney U test

### Figure 6. PF-10 score according to therapeutic success – Full Analysis Set (FAS)

[line/bar charts of the mean/median PF-10 at the baseline visit (visit 1) and the visit after 6 weeks (visit 2) according to therapeutic success]

### Patient's general condition - PGE score

A descriptive analysis of the PGE score at the baseline visit (visit 1) and the visit after 6 weeks (visit 2) will be conducted in this section, to assess the patient's general condition according to the investigator, using an 8-point ordinal scale from 1 (very poor) to 8 (excellent).

| | neral condition of the pa<br>e baseline visit and after<br>Analysis S | 6 weeks in complete | • |
|---|---|---|---|
| | Baseline 6 weeks P <sup>1</sup> (Visit 1) (Visit 2) | | |
| PGE score n (%) | | | |
| 1 | | | |
| 2 | | | |

OTIVACTO (1237.58) - SAP

Date: 18/02/2019 (Final Version 2.0) CONFIDENTIAL Página 40 de 68

| Table 24. | General condition of the patient – PGE score as assessed by the |
|---|---|
| physiciar | at the baseline visit and after 6 weeks in completed patients – Full |
| | Analysis Set (FAS) |

| | Baseline<br>(Visit 1) | 6 weeks<br>(Visit 2) | P <sup>1</sup> |
|---|---|---|---|
| 3 | | | |
| 4 | | | |
| 5 | | | |
| 6 | | | |
| 7 | | | |
| 8 | | | |
| Pooled PGE Score n (%) | | | |
| Poor (1-2) | | | |
| Satisfactory (3-4) | | | |
| Good (5-6) | | | |
| Excellent (7-8) | | | |

<sup>&</sup>lt;sup>1</sup> McNemar test

Figure 7. Patient's general condition –PGE score as assessed by the physician – Full Analysis Set (FAS)

[bar chart of PGE score at the baseline visit (visit 1) and the visit after 6 weeks (visit 2)]

[bar chart of pooled PGE score at the baseline visit (visit 1) and the visit after 6 weeks (visit 2)]

### Patient satisfaction with Spiolto® Respimat®

A descriptive analysis of patient satisfaction with Spiolto® Respimat® after 6 weeks of treatment (visit 2) will be conducted in this section, using a 7-point ordinal scale, from 1 (very satisfied) to 7 (very dissatisfied).

| Table 25.<br>trea | Patient satisfaction with Spiolto® Respima<br>tment (visit 2) in completed patients - Full Ar | |
|---|---|---|
| | | Total<br>n (%) |
| Patient overall satisfac<br>Respimat® treatment | tion with inhalation with the Spiolto® | |
| Very unsatisfied | | |
| Unsatisfied | | |
| Rather unsatisfied | | |
| Neither satisfied, no | r unsatisfied | |
| Rather satisfied | | |
| Satisfied | | |
| Very satisfied | | |

| Table 25. | Patient sati | sfaction with S | spiolto® Respima | t <sup>®</sup> after 6 weeks of |
|---|---|---|---|---|
| treat | ment (visit 2) | in completed i | patients - Full An | alysis Set (FAS) |

Total n (%)

## Patients satisfaction with inhaling from Respimat® device?

Very unsatisfied

Unsatisfied

Rather unsatisfied

Neither satisfied, nor unsatisfied

Rather satisfied

Satisfied

Very satisfied

# Patients satisfaction with haling of the Respimat® inhalation device?

Very unsatisfied

Unsatisfied

Rather unsatisfied

Neither satisfied, nor unsatisfied

Rather satisfied

Satisfied

Very satisfied

Figure 8. Patient satisfaction with Spiolto® Respimat® - Full Analysis Set (FAS)

[cumulative bar charts for the three items ]

OTIVACTO (1237.58) - SAP

Date: 18/02/2019 (Final Version 2.0) CONFIDENTIAL Página 42 de 68

<sup>&</sup>lt;sup>1</sup>Chi-square test/Fisher's exact test

# 6.5. SAFETY ANALYSIS (TS)

This section will describe the data related to suspected adverse reactions linked to Spiolto® Respimat® (serious or non-serious) and/or adverse events not related to Spiolto® Respimat®, but with a fatal outcome, reported by patients during the course of the study.

Pregnancies will also be indicated, at the start and at the end of the study. The sample analysed will be the **Treated Set** (n=xxx, see Table 4).

| Table 26. | Adverse events (AE) overall summary - Treated Set (TS) |
|---|---|
| | Total |
| | n (%) |
| Number of patients | |
| Patients with investiga | ator defined drug-related AE |
| Patients with invest leading to discontinua | igator defined drug-related AE<br>tion of trial drug |
| Patients with serious A | ΛΕ |
| Mortal | |
| Life-threatening | |
| Incapacity | |
| Hospitalisation | |
| Prolongation of hosp | italisation |
| Congenital anomaly | |
| Patients with serious A | AE leading to discontinuation |
| Patients with serious | drug-related AE |

## 6.5.1. Adverse events

| | Table 27. | AE according to MedDRA-SOC and PT - Treated Set (TS) | |
|---|---|---|---|
| | | Patients | Events |
| | | n (%) | n (%) |
| Presence of | AE during the | e study n (%) | |
| SOC 1 | | | |
| PT1 | | | |
| PT2 | | | |
| ••• | | | |
| SOC 2 | | | |
| PT1 | | | |

| | Table 27. | AE according to MedDRA-SOC and PT - Treated Set (TS) | |
|---|---|---|---|
| | | Patients | Events |
| | | n (%) | n (%) |
| PT2 | | | |

# 6.5.2. Drug-related adverse events

| Table 28. | Summary Drug-related adverse events - Treated Set (TS) |
|---|---|
| | Events |
| | n (%) |
| Total drug-related adv | verse events |
| Serious Drug-related a | dverse event |
| Non-Serious drug-rela | ted adverse event |

| | Table 29. | Serious Drug-related adverse events - Treated Set (TS) |
|---|---|---|
| | | Events |
| | | n (%) |
| Total Seri | ous drug-rela | ted adverse events |
| Description | on | |
| SOC 1 | | |
| PT1 | | |
| PT2 | | |
| ••• | | |
| SOC 2 | | |
| PT1 | | |
| PT2 | | |
| ••• | | |

| Table 30. | Non-Serious Drug-related adverse events - Treated Set (TS) |
|---|---|
| | Events |
| | n (%) |
| Total Non-Serious d | rug-related adverse events |
| Description | |
| SOC 1 | |
| PT1 | |



| Table 31. | Outcome Drug-related adverse events - Treated Set (TS) |
|---|---|
| | Events |
| | n (%) |
| Total drug-related adv | verse events |
| Outcome | |
| Recovered/resolved | |
| Not recovered/resolved | |
| Recovered/resolved with sequelae | |
| Exitus | |
| Unknown | |

## 6.5.3. Serious Adverse Events

| Table 32. | Characteristics of Serious adverse events - Treated Set (TS) |
|---|---|
| | Total |
| | n (%) |
| Total Serious adverse | events |
| Description | |
| SOC 1 | |
| PT 1 | |
| SOC 2 | |

Date: 18/02/2019 (Final Version 2.0) CONFIDENTIAL Página 45 de 68

### 6.5.4. Pregnancy

| Table 33. | Patient pregnant at AE - Treated Set (TS) |
|---------------------|-------------------------------------------|
| | n (%) |
| Total Patient at AE | |
| Yes | |
| No | |
| Not applicable | |

All AEs reported in the study, together with the provided characteristics of intensity, severity, treatment administered to treat the AR, action taken, causal relationship with study treatment and outcome will be listed in the ANNEX 7. REPORTED ADVERSE EVENTS.

Date: 18/02/2019 (Final Version 2.0)













### 7. REFERENCES

- 1 Vilagut G, et al. El Cuestionario de Salud SF-36 español: una década de experiencia y nuevos desarrollos [The Spanish version of the Short Form 36 Health Survey: a decade of experience and new developments]. Gac Sanit. 2005;19(2):135-50
- 2 Global Initiative for Chronic Obstructive Lung Disease (GOLD). Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease (updated 2014). http://www.goldcopd.org/uploads/users/files/GOLD\_Report\_2014.pdf (access date: 22 January 2014); Global Initiative for Chronic Obstructive Lung Disease (GOLD) (2014)
- 3 Global Initiative for Chronic Obstructive Lung Disease (GOLD). Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease (updated 2017). https://goldcopd.org/gold-2017-global-strategy-diagnosis-management-prevention-copd/(access date: 15 May 2017) Global Initiative for Chronic Obstructive Lung Disease (GOLD) (2017)

Date: 18/02/2019 (Final Version 2.0) CONFIDENTIAL Page 54 of 68

# 8. ANNEX

# 8.1. ANNEX 1. DB DEBUGGING

The DB debugging process, which is established in the Data Management Plan (DMP) will be described in this annex.

The description of debugging and/or variables generated during the data analysis process will also be described.

| | Table 48. Validation during data entry: Selection criteria | | |
|---|---|---|---|
| , | | Can be validated | |
| | | | No |
| | | | No |

[Note, if applicable]

| | | Table 49 | 9. Debugging | Debugging performed during the statistical analysis | |
|---|---|---|---|---|---|
| Patient | Visit | Variable | Data block | Inconsistency in DB | Action taken |

[Note, if applicable]

| | Table 50. | New variables created for the preparation of the results report | |
|---|---|---|---|
| New variable | | Data block | Description |

# 8.2. ANNEX 2. DETAILS OF THE NON-ASSESSABLE PATIENTS

This section will include the list of non-assessable patients for this study:

| | Table 51. | Description of the TS non-assessable patients | |
|---|---|---|---|
| Patient<br>No. | Inclusion criterion 1 | Informed consent date | Patient with no data on treatment<br>with Spiolto® Respimat® |

| Table 52. Description of the FAS non-assessable patients | | | | | | |
|---|---|---|---|---|---|---|
| Patient<br>No. | Inclusion<br>criterion<br>1 | Informed<br>consent<br>date | Patient with no<br>data on<br>treatment with<br>Spiolto®<br>Respimat® | Patients<br>with PF-10<br>assessable<br>at baseline<br>visit only | Patients with PF-10 assessable at visit after 6 weeks only | Patients without<br>PF-10 assessable<br>at baseline visit<br>and at visit after 6<br>weeks |

# 8.3. ANNEX 3. RECORDED CONCOMITANT DISEASES

Concomitant diseases recorded throughout the study, according to Table 12 (concomitant diseases at the baseline visit); and Table 18 (new concomitant diseases after 6 weeks) will be listed in the following tables.

| Table 53. | Concomitant disease | s at baseline | visit (visit 1) – Tre | eated Set (TS) |
|---|---|---|---|---|
| | | Total <sup>1</sup> | Total with CDs <sup>2</sup> | Ongoing <sup>2</sup> |
| Does the patient pres | | | | |
| Yes | | | | |
| No | | | | |
| Cardiovascular diseas | <b>e</b> n (%) | | | |
| Yes | | | | |
| No | | | | |
| Type of cardiovascular (diagnosis) <sup>3</sup> | disease | | | |
| Diagnosis 1 | | | | |
| Diagnosis | | | | |
| Diabetes mellitus n (% | 6) | | | |
| Yes | | | | |
| No | | | | |
| Musculoskeletal disor | ders n (%) | | | |
| Yes | | | | |
| No | | | | |
| Type of musculoskelet (diagnosis) <sup>4</sup> | al disorder | | | |
| Diagnosis 1 | | | | |
| Diagnosis | | | | |
| Kidney diseases n (%) | | | | |
| Yes | | | | |
| No | | | | |
| Type of kidney disease | (diagnosis) <sup>5</sup> | | | |
| Diagnosis 1 | | | | |
| Diagnosis | | | | |
| Liver diseases n (%) | | | | |
| Yes | | | | |
| No | | | | |
| Type of liver disease (d | liagnosis) <sup>6</sup> | | | |
| Diagnosis 1 | | | | |
| Diagnosis | | | | |

| | Table 53. | Concomitant diseases a | t baseline | visit (visit 1) – Tro | eated Set (TS) |
|---|---|---|---|---|---|
| | | | Total <sup>1</sup> | Total with CDs <sup>2</sup> | Ongoing <sup>2</sup> |
| Osteo | oorosis n (%) | | | | |
| Yes | | | | | |
| No | | | | | |
| Gastro | -oesophageal | reflux (GOR) n (%) | | | |
| Yes | | | | | |
| No | | | | | |
| Lung c | ancer n (%) | | | | |
| Yes | | | | | |
| No | | | | | |
| Other | n (%) | | | | |
| Yes | | | | | |
| No | | | | | |
| Туре о | f liver disease | (diagnosis) <sup>7</sup> | | | |
| Diagno | osis 1 | | | | |
| Diagno | osis | | | | |

Note: Concomitant disease (CD). A patient could have more than one CD

<sup>&</sup>lt;sup>7</sup> In the event of other concomitant diseases (n=xx)

| Table 54. | Dura | tion of co | ncomit | ant disea | ses at basel | ine visit (month | ns) ) – Treat | ted Set (TS) |
|---|---|---|---|---|---|---|---|---|
| | n | mean | SD | (95%<br>CI) | Median | [P25-P75] | Min | Max |
| Cardiovascular disease | | | | | | | | |
| Diagnosis 1 | | | | | | | | |
| Diagnosis | | | | | | | | |
| Diabetes mellitus | | | | | | | | |
| Musculoskeletal disorders | | | | | | | | |
| Diagnosis 1 | | | | | | | | |
| Diagnosis | | | | | | | | |
| Kidney diseases | | | | | | | | |
| Diagnosis 1 | | | | | | | | |
| Diagnosis | | | | | | | | |
| Liver diseases | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Of the total number of treated patients (n=xx)

<sup>&</sup>lt;sup>2</sup> Of the total number of patients with CDs (n=xx)

<sup>&</sup>lt;sup>3</sup> In the event of cardiovascular disease (n=xx)

<sup>&</sup>lt;sup>4</sup> In the event of osteoporosis (n=xx)

<sup>&</sup>lt;sup>5</sup> In the event of kidney diseases (n=xx)

<sup>&</sup>lt;sup>6</sup> In the event of liver diseases (n=xx)

| Diagnosis 1<br>Diagnosis |
|----------------------------------------|
| Osteoporosis |
| Gastro-<br>oesophageal<br>reflux (GOR) |
| Lung cancer |
| Other |
| Diagnosis 1 |
| Diagnosis |

Note: n according to each of the concomitant diseases

| Table 55. | New concomitant disease | | | |
|---|---|---|---|---|
| | | Total <sup>1</sup> | Total with<br>new CD <sup>2</sup> | Ongoing <sup>2</sup> |
| | eve any new concomitant ect to those of the last | | | |
| Yes | | | | |
| No | | | | |
| Cardiovascular dise | <b>ase</b> n (%) | | | |
| Yes | | | | |
| No | | | | |
| Diagnosis 1 | lar disease (diagnosis)³ | | | |
| Diagnosis | (0/) | | | |
| <b>Diabetes mellitus</b> n<br>Yes | (70) | | | |
| No | | | | |
| Musculoskeletal dis | sorders n (%) | | | |
| Yes | | | | |
| No | | | | |
| Type of musculoske<br>Diagnosis 1 | letal disorder (diagnosis) <sup>4</sup> | | | |
| Diagnosis | | | | |
| Kidney diseases n (9 | %) | | | |
| Yes | | | | |
| No | | | | |
| Type of kidney dised | ıse (diagnosis) <sup>5</sup> | | | |
| Diagnosis 1 | | | | |
| Diagnosis | | | | |

| Table 55. New concomitant diseases after 6 weeks (visit 2) ) – Treated Set (T | | | | |
|---|---|---|---|---|
| | Tota | al <sup>1</sup> | Total with new CD <sup>2</sup> | Ongoing <sup>2</sup> |
| Liver diseases n (%) | | | | |
| Yes | | | | |
| No | | | | |
| Type of liver disease | (diagnosis) <sup>6</sup> | | | |
| Diagnosis 1 | | | | |
| Diagnosis | | | | |
| Osteoporosis n (%) | | | | |
| Yes | | | | |
| No | | | | |
| Gastro-oesophageal | reflux (GOR) n (%) | | | |
| Yes | | | | |
| No | | | | |
| Lung cancer n (%) | | | | |
| Yes | | | | |
| No | | | | |
| Other n (%) | | | | |
| Yes | | | | |
| No | | | | |
| Type of liver disease | (diagnosis) <sup>7</sup> | | | |
| Diagnosis 1 | | | | |
| Diagnosis | | | | |

Note: Concomitant disease (CD). A patient could have more than one CD

<sup>&</sup>lt;sup>7</sup> In the event of other concomitant diseases (n=xx)

| Table 56. | Dura | Duration of new concomitant diseases after 6 weeks (months) – Treated Set (TS) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | n | mean | SD | (95% CI) | Median | [P25-P75] | Min | Max |
| Cardiovascular disease | | | | | | | | |
| Diagnosis 1 | | | | | | | | |
| Diagnosis | | | | | | | | |
| Diabetes mellitus | | | | | | | | |
| Musculoskeletal<br>disorders<br>Diagnosis 1 | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Of the total number of treated patients (n=xx)

<sup>&</sup>lt;sup>2</sup> Of the total number of patients with new CD (n=xx)

<sup>&</sup>lt;sup>3</sup> In the event of cardiovascular disease (n=xx)

<sup>&</sup>lt;sup>4</sup> In the event of osteoporosis (n=xx)

<sup>&</sup>lt;sup>5</sup> In the event of kidney diseases (n=xx)

<sup>&</sup>lt;sup>6</sup> In the event of liver diseases (n=xx)

| Table 56. | Dura | tion of ne | w con | comitant dis<br>Set (T | | 6 weeks (mo | nths) – 1 | reated |
|---|---|---|---|---|---|---|---|---|
| | n | mean | SD | (95% CI) | Median | [P25-P75] | Min | Max |
| Diagnosis | | | | | | | | |
| Kidney diseases | | | | | | | | |
| Diagnosis 1 | | | | | | | | |
| Diagnosis | | | | | | | | |
| Liver diseases | | | | | | | | |
| Diagnosis 1 | | | | | | | | |
| Diagnosis | | | | | | | | |
| Osteoporosis | | | | | | | | |
| Gastro-<br>oesophageal<br>reflux (GOR) | | | | | | | | |
| Lung cancer | | | | | | | | |
| Other | | | | | | | | |
| Diagnosis 1 | | | | | | | | |
| Diagnosis | | | | | | | | |

Note: n according to each of the concomitant diseases

### 8.4. ANNEX 4. CONCOMITANT MEDICATION

Concomitant medications administered throughout the study, according to Table 13 (concomitant medication at the baseline visit) and Table 19 (additional concomitant medication after 6 weeks) will be listed in the following tables.

| Table 57. Concomitant medication | on at baseline v | isit (visit 1) – Treat | ed Set (TS) |
|---|---|---|---|
| | Total <sup>1</sup> | Total with CM <sup>2</sup> | Ongoing <sup>2</sup> |
| Is the patient receiving any concomitant medication? n (%) | | | |
| Yes | | | |
| No | | | |
| Indication of the concomitant medication - Yes n (%) | | | |
| Indication 1 | | | |
| XXXXX | | | |
| XXXXX | | | |
| Indication 2 | | | |
| XXXXX | | | |
| XXXXX | | | |
| Indication 3 | | | |
| XXXXX | | | |
| XXXXX | | | |

Note: Concomitant medication (CM). The same patient could have more than one CM

| Table 58. | Duration of o | oncomita | nt me | dication at b | oaseline vis | it (months) – | Treated | Set (TS) |
|---|---|---|---|---|---|---|---|---|
| | n | mean | SD | (95% CI) | Median | [P25-P75] | Min | Max |
| Indication 1 | | | | | | | | |
| xxxx | | | | | | | | |
| xxxx | | | | | | | | |
| Indication 2 | | | | | | | | |
| xxxx | | | | | | | | |
| xxxx | | | | | | | | |
| Indication 3 | | | | | | | | |
| xxxx | | | | | | | | |
| xxxx | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Of the total number of treated patients (n=xx)

<sup>&</sup>lt;sup>2</sup> Of the total number of patients with CM (n=xx)

| Table 58. | Duration of o | Duration of concomitant medication at baseline visit (months) – Treated Set (TS) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | n | mean | SD | (95% CI) | Median | [P25-P75] | Min | Max |

Note: n according to each of the concomitant medications

| Table 59. Additional cond | Additional concomitant medication after 6 weeks (visit 2) – Treated Set (TS) | | | |
|---|---|---|---|---|
| | | Total <sup>1</sup> | Total with CM <sup>2</sup> | Ongoing <sup>2</sup> |
| Is the patient receiving any additional medication? $n (\%)$ | concomitant | | | |
| Yes | | | | |
| No | | | | |
| Indication of the additional concomitan Yes n (%) | t medication - | | | |
| Indication 1 | | | | |
| xxxxx | | | | |
| xxxxx | | | | |
| Indication 2 | | | | |
| xxxxx | | | | |
| XXXXX | | | | |
| Indication 3 | | | | |
| XXXXX | | | | |
| XXXXX | | | | |

Note: Concomitant medication (CM). The same patient could have more than one CM

| Table 60. | Duration | Duration (months) of the additional concomitant medication after 6 weeks (visit 2) – Treated Set (TS) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | n | mean | SD | (95%<br>CI) | Median | [P25-<br>P75] | Min | Max |
| Indication 1 | | | | | | | | |
| xxxx | | | | | | | | |
| XXXX | | | | | | | | |
| Indication 2 | | | | | | | | |
| xxxx | | | | | | | | |
| XXXX | | | | | | | | |
| Indication 3 | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Of the total number of treated patients (n=xx)

 $<sup>^{2}</sup>$  Of the total number of patients with CM (n=xx)

| Table 60. | Duration | Duration (months) of the additional concomitant medication after 6 weeks (visit 2) – Treated Set (TS) | |
|---|---|---|---|
| | n mean SD (95% Median [P25-<br>CI) Median P75] | | Max |
| xxxx | | | |
| xxxx | | | |

Note: n according to each of the concomitant medications

# 8.5. ANNEX 5. PREVIOUS TREATMENT FOR COPD

Previous treatments for COPD (in the 6 months prior to the baseline visit), as well as the duration, according to Table 14 (medication) will be specified in the following tables.

| Table 61. Treatment for COPD in the 6 m (visit 1) - Active Substance | • | oaseline visit |
|---|---|---|
| Total <sup>1</sup> | Total COPD <sup>2</sup> | Ongoing <sup>2</sup> |
| Has the patient received treatment for COPD in the previous 6 months? n (%) | | |
| Yes<br>No | | |
| Specify treatment for COPD - Yes n (%) | | |
| SAMA | | |
| Active substance 1 (units) | | |
| Active substance (units) | | |
| SABA | | |
| Active substance 1 (units) | | |
| Active substance (units) | | |
| LAMA | | |
| Active substance 1 (units) | | |
| Active substance (units) | | |
| LABA | | |
| Active substance 1 (units) | | |
| Active substance (units) | | |
| ICS | | |
| Active substance 1 (units) | | |
| Active substance (units) | | |
| LAMA/LABA n (%) | | |
| Active substance 1 (units) | | |
| Active substance (units) | | |
| LABA/ICS n (%) | | |
| Active substance 1 (units) | | |
| Active substance (units) | | |
| Other | | |
| Active substance 1 (units) | | |
| Active substance (units) | | |

| Table 62. | | Duration of treatment for COPD in the 6 months prior to the baseli visit (visit 1) - Active substance – Treated Set (TS) | | | | | |
|---|---|---|---|---|---|---|---|
| | n | mean | SD | (95% CI) | Median | [P25-P75] | 25-P75] Min |
| SAMA | | | | | | | |
| Active substance 1 | | | | | | | |
| (units) | | | | | | | |
| Active substance | | | | | | | |
| (units) | | | | | | | |
| SABA | | | | | | | |
| Active substance 1 | | | | | | | |
| (units) | | | | | | | |
| Active substance | | | | | | | |
| (units) | | | | | | | |
| LAMA | | | | | | | |
| Active substance 1 (units) | | | | | | | |
| (units)<br>Active substance | | | | | | | |
| (units) | | | | | | | |
| LABA | | | | | | | |
| Active substance 1 | | | | | | | |
| (units) | | | | | | | |
| Active substance | | | | | | | |
| (units) | | | | | | | |
| ICS | | | | | | | |
| Active substance 1 | | | | | | | |
| (units) | | | | | | | |
| Active substance | | | | | | | |
| (units) | | | | | | | |
| LAMA/LABA | | | | | | | |
| Active substance 1 | | | | | | | |
| (units) | | | | | | | |
| Active substance | | | | | | | |
| (units) LABA/ICS | | | | | | | |
| Active substance 1 | | | | | | | |
| (units) | | | | | | | |
| Active substance | | | | | | | |
| (units) | | | | | | | |
| Other | | | | | | | |
| Active substance 1 | | | | | | | |
| (units) | | | | | | | |
| Active substance | | | | | | | |
| (units) | | | | | | | |

Note: n according to each of the treatments for COPD

### 8.6. ANNEX 6. CURRENT TREATMENT FOR COPD

This annex will specify the current concomitant treatment (active substance) for COPD (SABA, ICS-Table 15), as well as the treatment dose.

| Table 63. | Current treatment for COPD (visit 1) – Treated Set (TS) |
|---|---|
| | Total |
| Is the patient going to re<br>COPD? n (%) | eceive other inhaled treatments for |
| Yes | |
| No | |
| Other inhaled treatment | s for COPD¹n (%) |
| SABA | |
| Active substance 1 (u | nits) |
| Active substance (u | nits) |
| ICS | |
| Active substance 1 (u | nits) |
| Active substance (u | nits) |

<sup>&</sup>lt;sup>1</sup> If the patient has received any other treatment for COPD (n=xx)

| | Table 64. | Current treatment for COPD (visit 2) – Treated Set (TS) |
|---|---|---|
| | | Total |
| Other inhal | ed treatment | s for COPD¹ n (%) |
| SABA | | |
| Active su | ubstance 1 (ur | nits) |
| Active su | ubstance (u | nits) |
| ICS | | |
| Active su | ubstance 1 (ur | nits) |
| Active su | ubstance (u | nits) |

<sup>&</sup>lt;sup>1</sup> If the patient has changed his/her concomitant medication for COPD (n=xx)

Date: 18/02/2019 (Final Version 2.0) CONFIDENTIAL Página 67 de 68

### 8.7. ANNEX 7. REPORTED ADVERSE EVENTS

This section will include the list of patients with reported AEs, , detailing the characteristics provided in terms of severity, reasonable causal relationship with the study drug (AR), action taken and outcome. In addition, the patient's gender and age will be specified.

| | Table 65. Individualised description of the adverse events under study – Treated Set (TS) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient code | Gender | Age | System organ class | Preferred<br>term | Reported term | Start<br>date | End date<br>(or<br>ongoing) | Intensity | Severity | Type of severity | Reasonable<br>relationship with<br>the study drug<br>(AR) | Action<br>taken | Outcome |

System organ class / Preferred term: Description of the adverse reaction according to SOC and PT of the MedDRA; Reported term: Description of the adverse reaction according to the investigator's description

| Table 66. Individualised description of the serious adverse events under study – Treated Set (TS) | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient code | Gender | Age | System organ class | Preferred<br>term | Reported<br>term | Start<br>date | End date<br>(or<br>ongoing) | Intensity | Severity | Type of severity | Reasonable<br>relationship with<br>the study drug<br>(AR) | Action<br>taken | Outcome |

System organ class / Preferred term: Description of the adverse reaction according to SOC and PT of the MedDRA; Reported term: Description of the adverse reaction according to the investigator's description